CLINICAL TRIAL: NCT04768361
Title: Behavioral Activation for Major Depressive Disorder: Comparison Between Protocols With and Without Mindfulness
Brief Title: Behavioral Activation for Major Depression With and Without Mindfulness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Miguel Servet (Other)
Responsible Party: Principal Investigator, Javier Garcia Campayo, Principal investigator, Hospital Miguel Servet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BA11.2019
Record Dates: First submitted 2019-11-11; First posted 2021-02-24 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Major Depressive Disorder
Keywords: Behavioral Activation; Mindfulness; Major depressive disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Activation without Mindfulness (Experimental): Program with 8 face to face sessions (115 minutes/session) in groups of 15-18 people. This program was adapted from BA proponents and excludes terms and interventions from Third Generation Therapies.
  Interventions: Behavioral: Behavioral Activation without Mindfulness
- Behavioral Activation with Mindfulness (Experimental): Program with 8 face to face sessions (115 minutes/session) in groups of 15-18 people. This program was adapted from BA proponents and include mindfulness practices.
  Interventions: Behavioral: Behavioral Activation with Mindfulness

INTERVENTIONS:
Behavioral: Behavioral Activation without Mindfulness — "Behavioral Activation without Mindfulness" includes functional analysis as key to defining out-of-session and activation strategies as central to mood change.
  Arms: Behavioral Activation without Mindfulness
Behavioral: Behavioral Activation with Mindfulness — "Behavioral Activation with Mindfulness" includes functional analysis as key to defining out-of-session and activation strategies and mindfulness as central to mood change.
  Arms: Behavioral Activation with Mindfulness

SUMMARY:
The objective of the study is to compare, in individuals who meet the diagnostic criteria for major depression, the effects of Behavioral Activation (BA) strictly behavioral with a BA protocol that includes mindfulness practices. The secondary objectives are: a) to verify if the changes in the level of depressive symptoms found after the treatment will be kept during the follow-up in both groups; b) evaluate the possible moderating role of baseline depression levels on the effectiveness of interventions; c) evaluate relapse rates after treatment; and d) test a BA protocol as a single treatment. The primary hypothesis is that BA protocol with mindfulness practices is superior to BA without mindfulness practices.

DETAILED DESCRIPTION:
Depression, according to the Word Health Organization, is the leading cause of disability in the world, often leading to a decrease in productivity and the departure from work activities, which generates economic impacts to the own health system. Between 2005 and 2015, an increase of almost 20% was identified in cases of depression worldwide. The impact of the disease on the world economy between 2011 and 2030 is expected at US $ 5,36 billion.

Behavioral Activation (BA) and interventions with mindfulness are recognized as effective for depression. On the other hand, as currently the BA is complemented with strategies of the Third Generation Therapies, including mindfulness, no study has compared a protocol strictly behavioral with any treatment and there is also insufficient data to affirm if the BA has better benefits than interventions that include or are based on mindfulness or vice versa.

The aim of this study is is to compare, in individuals who meet the diagnostic criteria for major depression, the effects of BA strictly behavioral with a BA protocol that includes mindfulness practices. The two intervention are face to face, in group (8 weeks), by a randomized controlled trial (RCT). Our main hypothesis is that la intervencion BA with mindfulness practices will be more efficacious to improve the symptomatology depressive, compared to a group with only BA the end of treatment. 150 participants diagnosed with depression will participate in the RCT.

ELIGIBILITY:
Inclusion Criteria:

* Be older than 18 years of age,
* To meet current DSM-5 criteria for major depression
* Be willing to participate in the study
* Be able to understand and read Spanish.

Exclusion Criteria:

* Not being able to read and write;
* Psychiatric conditions present that may affect study participation: schizophrenia, substance abuse, bipolar disorder, eating disorders, obsessive-compulsive disorder, social phobia, self-injurious behavior without suicidal intent;
* Be in psychotherapy;
* Have participated in three sessions of behavioral therapy and / or cognitive therapy;
* Have regular practice in any type of meditation;
* Disagreement in maintaining the dose of psychotropic medications without changes during the session period, if in use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2021-04-27 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | Basilene
  Beck Depression Inventory (BDI-II): instrument of 21 fragmented items that assesses levels of depressive symptoms in adolescents and adults. Each statement is followed by four options that correspond to a number (0, 1, 2 and 3) so that the participant responds according to the option that best describes how they felt in the last two weeks, including the day of the application of the instrument. The score ranges from 0 to 63. The internal consistency (α) and the correlation (p) found in the original study was .93 and an investigation conducted in Spain the value of Alpha was .89.
Behavioral Activation | Basilene
  Behavioral Activation Scale for Depression - Long Form (BADS): instrument that identifies the levels of activation and avoidance with 25 elements which must be answered from a Likert scale of 0 ("disagree") to 6 ("Totally agree") considering the last week, including the day of application of the instrument. The internal consistency of the total scale obtained in a first study was .92 and with a population of Spanish obtained a similar value of .90.
Depressive symptoms | 8 weeks
  Beck Depression Inventory (BDI-II): instrument of 21 fragmented items that assesses levels of depressive symptoms in adolescents and adults. Each statement is followed by four options that correspond to a number (0, 1, 2 and 3) so that the participant responds according to the option that best describes how they felt in the last two weeks, including the day of the application of the instrument. The score ranges from 0 to 63. The internal consistency (α) and the correlation (p) found in the original study was .93 and an investigation conducted in Spain the value of Alpha was .89.
Behavioral Activation | 8 weeks
  Behavioral Activation Scale for Depression - Long Form (BADS): instrument that identifies the levels of activation and avoidance with 25 elements which must be answered from a Likert scale of 0 ("disagree") to 6 ("Totally agree") considering the last week, including the day of application of the instrument. The internal consistency of the total scale obtained in a first study was .92 and with a population of Spanish obtained a similar value of .90.
Depressive symptoms | 6 months follow up
  Beck Depression Inventory (BDI-II): instrument of 21 fragmented items that assesses levels of depressive symptoms in adolescents and adults. Each statement is followed by four options that correspond to a number (0, 1, 2 and 3) so that the participant responds according to the option that best describes how they felt in the last two weeks, including the day of the application of the instrument. The score ranges from 0 to 63. The internal consistency (α) and the correlation (p) found in the original study was .93 and an investigation conducted in Spain the value of Alpha was .89.
Behavioral Activation | 6 months follow up
  Behavioral Activation Scale for Depression - Long Form (BADS): instrument that identifies the levels of activation and avoidance with 25 elements which must be answered from a Likert scale of 0 ("disagree") to 6 ("Totally agree") considering the last week, including the day of application of the instrument. The internal consistency of the total scale obtained in a first study was .92 and with a population of Spanish obtained a similar value of .90.

SECONDARY OUTCOMES:
Automatic Thought Questionnarie (ATQ) | Basilene
  Instrument consisting of 30 items that seeks to measure the frequency of negative thoughts related to depression. The participant must respond on the basis of the last week, including the day of application of instrument, the frequency of the thoughts using a Likert-type scale from 1 ("in absolute") to 5 ("al time"). The internal consistency found at the first validation was from .97 and the adaptation to Spanish found the values of .94 for negative self-concept, hopelessness .93, .87 for maladjustment and .85 for the self-disapproval.
Daily Activity Record (RAD) | Basilene
  Consists of a table for daily logging of activities performed by the individual, classifying the mood between 0 and 10. It may be 0 = "not depressed" and 10 "very depressed" or the other hand, 0 = "very depressed" and 10 = "not depressed"

OTHER OUTCOMES:
Five Facet Mindfulness Questionnaire (FFMQ) | Basilene
  Instrument contains 39 fragmented items into five factors (observing, describing, acting with awareness, nojudging and nonreactivity) that are answered from a Likert scale of 1 ("never" or "very rarely true") to 5 ("very often" or "always true"). The internal consistency (α) and the correlation (p) found in a first study was: observing = .83, describing = .91, acting with awareness = .87, non-judging = 0.87. and nonreactivity = .75. In the Spanish language was found: observing = .81, describing = .91, acting with awareness = .89, nojudging = 0.91. y nonreactivity = .80.
Automatic Thought Questionnarie (ATQ) | 8 weeks
  Instrument consisting of 30 items that seeks to measure the frequency of negative thoughts related to depression. The participant must respond on the basis of the last week, including the day of application of instrument, the frequency of the thoughts using a Likert-type scale from 1 ("in absolute") to 5 ("al time"). The internal consistency found at the first validation was from .97 and the adaptation to Spanish found the values of .94 for negative self-concept, hopelessness .93, .87 for maladjustment and .85 for the self-disapproval.
Daily Activity Record (RAD) | 8 weeks
  Consists of a table for daily logging of activities performed by the individual, classifying the mood between 0 and 10. It may be 0 = "not depressed" and 10 "very depressed" or the other hand, 0 = "very depressed" and 10 = "not depressed"
Five Facet Mindfulness Questionnaire (FFMQ) | 8 weeks
  Instrument contains 39 fragmented items into five factors (observing, describing, acting with awareness, nojudging and nonreactivity) that are answered from a Likert scale of 1 ("never" or "very rarely true") to 5 ("very often" or "always true"). The internal consistency (α) and the correlation (p) found in a first study was: observing = .83, describing = .91, acting with awareness = .87, non-judging = 0.87. and nonreactivity = .75. In the Spanish language was found: observing = .81, describing = .91, acting with awareness = .89, nojudging = 0.91. y nonreactivity = .80.
Automatic Thought Questionnarie (ATQ) | 6 months follow up
  Instrument consisting of 30 items that seeks to measure the frequency of negative thoughts related to depression. The participant must respond on the basis of the last week, including the day of application of instrument, the frequency of the thoughts using a Likert-type scale from 1 ("in absolute") to 5 ("al time"). The internal consistency found at the first validation was from .97 and the adaptation to Spanish found the values of .94 for negative self-concept, hopelessness .93, .87 for maladjustment and .85 for the self-disapproval.
Daily Activity Record (RAD) | 6 months follow up
  Consists of a table for daily logging of activities performed by the individual, classifying the mood between 0 and 10. It may be 0 = "not depressed" and 10 "very depressed" or the other hand, 0 = "very depressed" and 10 = "not depressed"
Five Facet Mindfulness Questionnaire (FFMQ) | 6 months follow up
  Instrument contains 39 fragmented items into five factors (observing, describing, acting with awareness, nojudging and nonreactivity) that are answered from a Likert scale of 1 ("never" or "very rarely true") to 5 ("very often" or "always true"). The internal consistency (α) and the correlation (p) found in a first study was: observing = .83, describing = .91, acting with awareness = .87, non-judging = 0.87. and nonreactivity = .75. In the Spanish language was found: observing = .81, describing = .91, acting with awareness = .89, nojudging = 0.91. y nonreactivity = .80.

CONTACTS AND LOCATIONS:
Overall Officials: Javier García-Campayo, Principal Investigator — Miguel Servet Hospital and University os Zaragoza, Spain
Locations (1):
- Department of Psychiatry. Miguel Servet University Hospital, Zaragoza, Spain

REFERENCES:
- [Background] Finning K, Richards DA, Moore L, Ekers D, McMillan D, Farrand PA, O'Mahen HA, Watkins ER, Wright KA, Fletcher E, Rhodes S, Woodhouse R, Wray F. Cost and outcome of behavioural activation versus cognitive behavioural therapy for depression (COBRA): a qualitative process evaluation. BMJ Open. 2017 Apr 13;7(4):e014161. doi: 10.1136/bmjopen-2016-014161. PMID 28408544
- [Background] Huguet A, Miller A, Kisely S, Rao S, Saadat N, McGrath PJ. A systematic review and meta-analysis on the efficacy of Internet-delivered behavioral activation. J Affect Disord. 2018 Aug 1;235:27-38. doi: 10.1016/j.jad.2018.02.073. Epub 2018 Mar 8. PMID 29649708
- [Background] Kanter JW, Baruch DE, Gaynor ST. Acceptance and commitment therapy and behavioral activation for the treatment of depression: description and comparison. Behav Anal. 2006 Fall;29(2):161-85. doi: 10.1007/BF03392129. PMID 22478462
- [Background] Parikh SV, Quilty LC, Ravitz P, Rosenbluth M, Pavlova B, Grigoriadis S, Velyvis V, Kennedy SH, Lam RW, MacQueen GM, Milev RV, Ravindran AV, Uher R; CANMAT Depression Work Group. Canadian Network for Mood and Anxiety Treatments (CANMAT) 2016 Clinical Guidelines for the Management of Adults with Major Depressive Disorder: Section 2. Psychological Treatments. Can J Psychiatry. 2016 Sep;61(9):524-39. doi: 10.1177/0706743716659418. Epub 2016 Aug 2. PMID 27486150
- [Background] Strauss C, Cavanagh K, Oliver A, Pettman D. Mindfulness-based interventions for people diagnosed with a current episode of an anxiety or depressive disorder: a meta-analysis of randomised controlled trials. PLoS One. 2014 Apr 24;9(4):e96110. doi: 10.1371/journal.pone.0096110. eCollection 2014. PMID 24763812
- See also: Mindful Nation UK (2015). Report by the Mindfulness All-Party Parliamentary Group (MAPPG) — https://www.themindfulnessinitiative.org/mindful-nation-report
- See also: UN health agency reports depression now 'leading cause of disability worldwide' — https://news.un.org/en/story/2017/02/552062-un-health-agency-reports-depression-now-leading-cause-disability-worldwide